CLINICAL TRIAL: NCT06629857
Title: Clinical Correlation of Alpha-Fetoprotein in Hepatocellular Carcinoma: a Cross-Sectional Study from Southeast Asia
Brief Title: A Cross Sectional Study Evaluating the Mean Levels of Alpha Fetoprotein in Patients of Hepatocellular Carcinoma and Its Correlates in Pakistan
Status: Completed | Type: Observational
Sponsor: Darul Sehat Hospital (Other)
Responsible Party: Principal Investigator, Maryam Abbasi, Principal investigator, Jinnah Sindh Medical University
Other Study IDs: M-000037/22
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma (HCC); Alpha-fetoprotein (AFP) levels; Liver cancer biomarkers; Tumor size and AFP correlation; Hepatitis B and C in liver cancer; Non-alcoholic steatohepatitis (NASH); AFP as a diagnostic tool; Liver tumor progression markers
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: HCC Patients with Elevated AFP Levels Description: This group includes patients diagnosed

SUMMARY:
This study aims to explore the levels of alpha-fetoprotein (AFP), a protein often elevated in liver cancer, in patients with hepatocellular carcinoma (HCC). The goal is to determine whether AFP levels vary based on the size of the liver tumor or other health conditions like hepatitis B, hepatitis C, and obesity. By analyzing data from 94 patients, the study seeks to identify factors that influence AFP levels, which may help in understanding liver cancer progression and improving diagnosis and treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 27 to 80 years.
* Diagnosed with hepatocellular carcinoma (HCC) within the last three months.
* Diagnosis confirmed by relevant investigations (e.g., imaging, liver biopsy).
* Able to provide informed consent.

Exclusion Criteria:

* Elevated alpha-fetoprotein levels due to tumors other than HCC.
* Presence of secondary liver metastases from other primary sites.
* Any significant comorbid conditions that could interfere with study assessments.
* Pregnancy or breastfeeding.

Ages: 27 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a total of 94 adult patients diagnosed with hepatocellular carcinoma (HCC) who are receiving care at Dar ul Sehat Hospital, Karachi, Pakistan. Participants will be recruited from outpatient, emergency, and inpatient departments. Eligible individuals will be aged between 27 to 80 years and must have been diagnosed with HCC within the last three months, confirmed by relevant investigations. The study aims to reflect a diverse population that includes various tumor sizes and underlying liver disease etiologies, such as hepatitis B, hepatitis C, non-alcoholic steatohepatitis, and cirrhosis. Patients will be excluded if they have elevated alpha-fetoprotein levels due to tumors other than HCC or have secondary liver metastases from other primary sites. This approach ensures that the findings are specific to HCC and its correlates, aiding in the assessment of AFP levels in this population.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Mean Alpha-Fetoprotein (AFP) Levels in HCC Patients | Baseline measurement at time of diagnosis.

SECONDARY OUTCOMES:
Correlation Between AFP Levels and Tumor Size | At baseline (upon diagnosis).

CONTACTS AND LOCATIONS:
Locations (1):
- Darul Sehat Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided